CLINICAL TRIAL: NCT03943433
Title: The Effect of Oxygen Concentration During Alveolar Recruitment on Absorption Atelectasis
Brief Title: Oxygen Concentration During Alveolar Recruitment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jae-Hyon Bahk, MD, PhD, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: JHBahk_AR
Record Dates: First submitted 2019-05-07; First posted 2019-05-09 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Atelectasis, Postoperative Pulmonary
Keywords: Absorption atelectasis; Lung sono; Oxygen concentration
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FiO2_1.0 (Active Comparator): Alveolar recruitment is performed with 100% oxygen concentration at specific time points.
  Interventions: Procedure: FiO2_1.0
- FiO2_0.4 (Experimental): Alveolar recruitment is performed with 40% oxygen concentration at specific time points.
  Interventions: Procedure: FiO2_0.4

INTERVENTIONS:
Procedure: FiO2_1.0 — Alveolar recruitment is performed with 100% oxygen concentration after general anesthesia induction, after position change to Trendelenburg, after position change to supine, and at the end of operation.
  Arms: FiO2_1.0
Procedure: FiO2_0.4 — Alveolar recruitment is performed with 40% oxygen concentration after general anesthesia induction, after position change to Trendelenburg, after position change to supine, and at the end of operation.
  Arms: FiO2_0.4

SUMMARY:
The purpose of this study is to investigate the effect of oxygen concentration during alveolar recruitment on absorption ateletasis.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing laparoscopic obstetric or colon surgery with Trendelenburg position

Exclusion Criteria:

* American Society of Anesthesiologists physical status IV or more
* Severe cardiovascular disease
* Severe chronic obstructive pulmonary disease, emphysema
* History of pneumothorax, bullae
* History of lung resection surgery
* Conversion to laparotomy
* Refusal to participate

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
Modified lung ultrasound score | Intraoperative (at the end of operation, before emergence)
  The score is calculated by adding up the 12 individual quadrant scores assessed using lung ultrasound. Each quadrant score ranges from 0 (minimal atelectasis)~3 (severe atelectasis), so the maximum total score is 36.

SECONDARY OUTCOMES:
Modified lung ultrasound score | Postoperative 30 minutes
  The score is calculated by adding up the 12 individual quadrant scores assessed using lung ultrasound. Each quadrant score ranges from 0 (minimal atelectasis)~3 (severe atelectasis), so the maximum total score is 36.
Intraoperative desaturation | Intraoperative
  Oxygen saturation by pulse oximetry <95%
Intraoperative partial pressure of arterial oxygen/fraction of inspired oxygen ratio | Intraoperative (20minutes after each recruitment)
  Partial pressure of arterial oxygen/fraction of inspired oxygen ratio
Postoperative partial pressure of arterial oxygen/fraction of inspired oxygen ratio | Postoperative 30 minutes
  Partial pressure of arterial oxygen/fraction of inspired oxygen ratio
Postoperative pulmonary complication | Postoperative 24 hours
  respiratory infection, respiratory failure, pleural effusion, atelectasis, pneumothorax, atelectasis, bronchospasm, aspiration pneumonitis

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Hyon Bahk, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim BR, Lee S, Bae H, Lee M, Bahk JH, Yoon S. Lung ultrasound score to determine the effect of fraction inspired oxygen during alveolar recruitment on absorption atelectasis in laparoscopic surgery: a randomized controlled trial. BMC Anesthesiol. 2020 Jul 18;20(1):173. doi: 10.1186/s12871-020-01090-y. PMID 32682397